CLINICAL TRIAL: NCT03064867
Title: Phase I/II Trial of Venetoclax in Combination With R-ICE (V+RICE) Chemotherapy for Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Venetoclax Plus R-ICE Chemotherapy for Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Molly Gallogly (Other)
Responsible Party: Sponsor-Investigator, Molly Gallogly, MD, PhD, Division of Hematology and Oncology, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2415
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Diffuse Large B-cell-lymphoma
Keywords: venetoclax; rituximab; ifosfamide; carboplatin; etoposide
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — venetoclax; Rituximab; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- V+RICE (Experimental): Venetoclax given in combination with R-ICE chemotherapy (rituximab, ifosfamide, carboplatin, and etoposide)
  Phase I part of this study is a 3 + 3 design, with 3 dose levels, a minimum of 6 participants (maximum of 18) will be required to identify the recommended phase 2 dose (RP2D).
  Phase II involvs two stages: In stage I, a total of 16 participants will be accrued. If there are 7 or fewer complete responses (CR), the study will be stopped. Otherwise, an additional 30 participants will be accrued in stage II.
  The maximum number of treatment cycles with V+RICE is three. Participants who achieve complete remission at the interim response assessment after 2 cycles may omit cycle 3 in order to proceed to subsequent consolidation therapy with autologous stem cell transplant (AHSCT).
  Participants will proceeed to other treatment including RICE, other chemotherapy, peripheral blood stemm cell collection, and ASCT per institutional guidelines.
  Interventions: Drug: Venetoclax; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Venetoclax — Beginning with 400mg daily on days 1-10 of cycle 1-3
  Phase I dose escalation scheme:
  Dose Level -2 (DL-2): 100 mg daily, days 1-10, cycle 1-3
  DL-1: 200 mg daily, days 1-10, cycle 1-3
  DL1: 400 mg daily, days 1-10, cycle 1-3
  DL2: 600 mg daily, days 1-10, cycle 1-3
  DL3: 800 mg daily, days 1-10, cycle 1-3
  Phase II: Given at a dose of 400mg daily for 5 days
Drug: Rituximab — Part of R-ICE treatment:
  Rituximab: 375 mg/m^2 intravenously (IV) on Day 1 of R-ICE every 21 days
  Other Names: Rituxan
Drug: Ifosfamide — Part of R-ICE treatment:
  Ifosfamide: 5,000 mg/m^2 mixed together with mesna at a dose of 5,000 mg/m^2 over 24 hours beginning on Day 2 and completing on Day 3 of each 21-day cycle
  Other Names: Ifex
Drug: Carboplatin — Part of R-ICE treatment:
  Carboplatin: At a dose corresponding to an AUC = 5 based on Cockcroft-Gault calculation of GFR using adjusted body weight. Carboplatin is given IV on the Day 2 of RICE of each 21 day cycle
  Other Names: Paraplatin
Drug: Etoposide — Part of R-ICE treatment:
  Etoposide: 100 mg/m2by IV daily on 3 consecutive days (Days 1-3) of each 21-day cycle
  Other Names: VP-16; VePesid

SUMMARY:
The purpose of this study is to determine the correct dose and safety of adding a new cancer drug, venetoclax, to a standard combination of chemotherapy drugs as a second treatment for relapsed/refractory DLBCL. In this study, venetoclax will be added to RICE (rituximab, ifosfamide, carboplatin, etoposide), a common set to cancer drugs used as a second line treatment for relapsed/refractory DLBCL.

Venetoclax, is a new targeted anti-cancer drug, which works by mimicking a particular protein produced by the tumor and interrupting its normal processes, ultimately causing the tumor cells to die. Adding venetoclax to the standard RICE regimen is believed to increase the chance of getting cancer into remission.

Venetoclax is experimental because it is not approved by the Food and Drug Administration (FDA) for the treatment of relapsed/refractory DLBCL. Venetoclax has been FDA approved for use in patients with chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
Primary Objective:

Establishment of safety of V+RICE in order to identify the recommended Phase II dose (RPD2)

Secondary Objectives:

1. Determine the overall response rate (ORR) of V+RICE relative to historical controls of RICE alone in r/r DLBCL.
2. Determine the proportion of patients who proceed to autologous stem cell transplantation after V+RICE relative to historical controls.
3. Describe the progression-free survival (PFS) and overall survival (OS) for patients treated with V + RICE who do and do not proceed to auto-Stem Cell Transplant, relative to historical controls.
4. Measure total number of peripheral blood stem cells collected in patients treated with V + RICE who proceed to stem cell mobilization/harvesting, compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of relapsed/refractory diffuse large B-cell lymphoma after prior rituximab and anthracycline-containing systemic treatment regimen such as R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone), R-EPOCH (rituximab, etoposide phosphate, prednisone, vincristine sulfate, cyclophosphamide, doxorubicin hydrochloride), R-HyperCVAD (rituximab, cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, dexamethasone) etc. A biopsy immediately before enrollment is not required.
* Subjects must have received no more than 2 prior systemic therapies for lymphoma. Prior therapy with systemic rituximab monotherapy or conventional chemotherapy (i.e. bendamustine, CVP (Cyclophosphamide, Vincristine Sulfate, Prednisone) or other) ± rituximab for indolent non-Hodgkin's lymphoma (NHL) ± maintenance/extended-use rituximab will count as 1 line of systemic therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2
* Subjects must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 8.0 g/dl
  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelet count ≥ 75,000/mcL
  * Total bilirubin ≤ 1.5 X the upper limit of normal (ULN) unless a known history of impaired bilirubin conjugation such as Gilbert's, for whom the maximum will be 2.5 ULN.
  * Aspartate transaminase (AST) (SGOT) ≤ 2.5 X institutional ULN
  * Alanine transaminase (ALT) (SGPT) ≤ 2.5 X institutional ULN
  * International normalized ratio (INR) ≤ 1.5 ×ULN
  * Patients must have a calculated serum creatinine clearance > 50 mL/min using Cockcroft-Gault calculation or based on 24-hour urine collection performed within 7 days prior to treatment.
* Specific guidelines will be followed regarding inclusion of relapsed/refractory DLBCL based on Hepatitis B serological testing as follow:

  * HBsAg negative, HBcAb negative, HBsAb negative patients are eligible.
  * HBsAg negative, HBcAb negative, HBsAb positive patients are eligible.
  * Patients who test positive for HBsAg are ineligible
  * Patients with HBsAg negative, but HBcAb positive (regardless of HBsAb status) should have a HBV DNA testing performed and protocol eligibility determined as follow:

    * If HBV DNA is positive, the subject is ineligible.
    * If HBV DNA is negative, the subject may be included but must undergo HBV DNA PCR testing monthly x 3 months beginning from the start of treatment
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 30 days after the last dose of venetoclax or 18 months after the last dose of rituximab, whichever is longer.

A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of rituximab. Men must refrain from donating sperm during this same period.

With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose of rituximab to avoid exposing the embryo.

Exclusion Criteria:

* Prior treatment toxicities have not resolved to ≤ Grade 2 according to NCI CTCAE Version 4.0 (except clinically insignificant toxicities such as alopecia).
* Subjects receiving any other investigational agents.
* Patients with active tumor lysis syndrome (TLS) either from laboratory or clinical changes.
* Patients with active central nervous system (CNS) disease defined as symptomatic meningeal lymphoma or known CNS parenchymal lymphoma.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to rituximab or other agents used in this study.
* Subjects with uncontrolled intercurrent illness .
* HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Venetoclax. In addition, these subjects are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated. HIV testing prior to enrollment is not required for screening but strongly encouraged for patients with no documented prior HIV assessment.
* Presence of positive test results for hepatitis B virus (HBV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) antibody.

  * Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation
  * Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable. These patients must be willing to undergo monthly DNA testing.
* Women who are pregnant or lactating
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Chemotherapy or radiation within 3 weeks of the first scheduled study treatment.
* Less than 2-year disease free from another primary malignancy (other than squamous or basal cell carcinoma of the skin, "in-situ" carcinoma of the cervix or breast, superficial bladder carcinoma, or previously treated localized prostate cancer with normal prostate specific antigen (PSA) levels). Patients who have had completed all anti-cancer treatment for another primary malignancy more than 2 years prior to screening are eligible if they are not considered to have a "currently active" malignancy based on having less than a 30% risk of relapse.
* Major surgery, other than diagnostic surgery, within 2 weeks.
* Medical condition requiring chronic use of high dose systemic corticosteroids (i.e., doses of prednisone higher than 10 mg/day or equivalent). Brief (<15 days) treatment with glucocorticoids (prednisone 100 mg by mouth daily, or equivalent) is acceptable.
* Known allergy to both xanthine oxidase inhibitors and rasburicase.
* Use of warfarin is prohibited. Anticoagulation with low-molecular weight heparin (i.e. enoxaparin) or direct thrombin inhibitors is permitted.
* The following concomitant medications are not allowed from 7 days prior to the first dose of study drug and during venetoclax administration: Strong CYP3A4 inhibitors including but not limited to fluconazole, ketoconazole, and clarithromycin or strong CYP3A4 inducers included but not limited to rifampin, carbamazepine.
* Receipt of live-virus vaccines within 28 days prior to the initiation of study treatment or need for live-virus vaccines at any time during study treatment.
* Concomitant medications that fall into the categories below could potentially lead to adverse reactions and should be considered with caution.

  * Moderate/Weak CYP3A inducers such as efavirenz and oxcarbazepine
  * CYP2C8 substrates such as thiazolidinediones (glitazones) and select statins (because of expected inhibition of the metabolism of CYP2C8 substrates) by venetoclax
  * CYP2C9 substrates such as tolbutamide (because of expected inhibition of the metabolism of CYP2C9 substrates by venetoclax. It is recommended to exclude CYP2C9 substrates with a narrow therapeutic index such as phenytoin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2023-08-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose | Up to 12 weeks
  A maximum of 18 patients can theoretically participate in the initial dose escalation with Retinoic and Lithium, based on 4 dose levels with a maximum of 6 patients at each dose level. At a true dose limiting toxicity rate of 20%, the chance of escalating to the next dose level is 71% and of establishing the lower dose level as maximum tolerated dose is 29%.

SECONDARY OUTCOMES:
Overall Response Rate | Up to 12 weeks
  number of patients with complete response or partial response as document in a positron emission tomography/ computerized tomography (PET/CT) scan and defined by the Revised Response Criteria for Malignant Lymphoma
Proportion of participants Proceeding to ASCT | Up to 12 weeks
  the number of patients with ASCT divided by the total number of patients
Progression Free Survival | Up to 12 weeks
  Average time disease did not progress as based on the Revised Response Criteria for Malignant Lymphoma up to 12 weeks
Overall Survival | Up to 12 weeks
  Average time participants are alive from starting treatment to death or 12 weeks, whichever comes first
Number of Peripheral Blood Stem Cells Collected | Up to 12 weeks
  Estimated through measurement of CD34+ cells/kg
Median Number of cluster of differentiation 34 (CD34+) Cells/kg | Up to 12 weeks
  Median value of CD34+ in cells/kg collected from patients

OTHER OUTCOMES:
Analysis for Myc | Up to 12 weeks
  Number of patients with mutant Myc regulatory gene
Analysis for Bcl-2 | Up to 12 weeks
  Number of patients with mutant B-cell lymphoma-2 genes

CONTACTS AND LOCATIONS:
Overall Officials: Molly Gallogly, MD PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Washington University School of Medicine, Siteman Cancer Center, St Louis, Missouri
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio